CLINICAL TRIAL: NCT06500078
Title: Effects of Intermittent Dietary Restriction on Cardiometabolic Risk in School-aged Children: A Randomized Controlled Trial
Brief Title: Effects of Intermittent Dietary Restriction on Cardiometabolic Risk in School-aged Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IM_Diet_2.0
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Syndrome, Metabolic
Keywords: Intermittent carbohydrate restriction; Intermittent calorie restriction; Cardiometabolic risk; Children
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent dietary restriction group (ILCD or ICR) (Experimental): Intermittent dietary restriction group will receive ILCD or ICR intervention. ILCD will be conducted as a carbohydrate intake restriction of ≤ 50 g/day for two consecutive or discontinuous days per week, and ICR will be conducted as a calorie intake restriction of 500-600 kcal/day for two consecutive or discontinuous days per week.
  Interventions: Behavioral: Intermittent dietary restriction; Behavioral: General health education
- Health education group (Active Comparator): Health education group will receive health education based on Chinese guidelines for school-aged children.
  Interventions: Behavioral: General health education

INTERVENTIONS:
Behavioral: Intermittent dietary restriction — Intermittent dietary restriction will include the ILCD and ICR, which will be self-administered interventions in daily lives. The ILCD intervention will ask participants to restrict carbohydrate intake to ≤ 50 g/d on two consecutive or discontinuous days per week. The ICR intervention will ask participants to restrict caloric intake to 600 kcal/d for boys and 500 kcal/d for girls on two consecutive or discontinuous days per week.
  At baseline, participants will receive face-to-face oral dietary instructions (e.g., principle of dietary restriction, sample menus, food list with macronutrients). Participants will receive the intervention booklets containing dietary advice and sample menus for diet according to the requirements of the dietary intervention.
  Participants will be required to record dietary and physical activity data on a regular basis. The total intervention duration will be 12 months, including a 3-month intervention phase and a 9-month self-maintenance phase.
  Arms: Intermittent dietary restriction group (ILCD or ICR)
Behavioral: General health education — General health education based on dietary and physical activity guidelines for Chinese children and adolescents, will regularly send offline and online promotional materials to participants.

SUMMARY:
This randomized trial aims to evaluate the health-promoting effects of intermittent dietary restrictions, including intermittent low-carbohydrate diet (ILCD) and calorie restriction (ICR), in school-aged children with cardiometabolic risk (CMR) compared with general health education based on dietary and physical activity guidelines for Chinese children.

DETAILED DESCRIPTION:
Childhood obesity comorbid with one or more CMR factors, including hyperglycemia, dyslipidemia, and hypertension, predicts an increased risk for developing cardiovascular disease in adulthood. Lifestyle interventions, including restricting dietary calorie intake and increasing physical activity, have been proposed as the first-line behavioral weight management approaches for pediatric obesity. Long-term adherence to daily dietary restriction is challenging for young populations because they are in a particular period of physical and psychological growth and lifestyle formation. Low-carbohydrate diet and ICR have shown effectiveness in improving cardiometabolic health in adults, however, the evidence supporting the effects of these diets in pediatric populations remains limited.

Eligible participants will be randomized to receive intermittent dietary restriction, including an ILCD (carbohydrate intake ≤ 50 g/d for two days per week) or an ICR (calorie intake is 500-600 kcal/d for two days per week), or general health education based on dietary and physical activity guidelines for Chinese children in daily life. The total study duration will be 12 months consisting of a 3-month intervention phase and a 9-month self-maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-18 years at baseline.
* At least one of the following cardio-metabolic abnormalities:

  1. Prediabetes (Impaired fasting glucose: 5.6 ≤ fasting blood glucose level ≤ 6.9 mmol/L; or Impaired glucose tolerance: 7.8 ≤ blood glucose level after 2 hours postprandial ≤ 11.0 mmol/L).
  2. Lipid abnormalities (High-density lipoprotein cholesterol ≤ 1.04 mmol/L; or Low-density lipoprotein cholesterol ≥ 3.37 mmol/L; or Triglycerides ≥ 1.70 mmol/L, or Total cholesterol ≥ 5.18 mmol/L).
  3. Elevated blood pressure (Systolic/diastolic blood pressure consistently higher than the 90th percentile for gender, age, and height; or systolic/diastolic blood pressure ≥ 120/80 mmHg).

Exclusion Criteria:

* Previously diagnosed with heart failure, severe malnutrition, immune deficiency, liver or kidney disease, cancer, or other diseases deemed unsuitable for participation.
* Had a history of bariatric surgery.
* Used weight loss pills or supplements in the last three months.
* Other situations unsuitable for participation.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reversal of at least one cardiometabolic abnormalities | At month 3 from baseline
  The primary outcome is a composite outcome that will be measured by combining multiple reverse outcomes of the following cardiometabolic abnormalities: (1) prediabetes; (2) lipid abnormalities; (3) elevated blood pressure. It is defined as occurring if any cardiometabolic abnormality has a reversal outcome at 3rd month of study phrase.
  Reversal of cardiometabolic abnormalities is defined as: at 3rd month of study phrase, at least one of the following status changed from abnormal at baseline to normal:
  i. Prediabetes; ii. Lipid abnormalities; iii. Elevated blood pressure.

SECONDARY OUTCOMES:
Number of participants with reversal of at least one cardiometabolic abnormalities | At month 12 from baseline
  It is a composite outcome that will be measured by combining multiple reverse outcomes of the following cardiometabolic abnormalities: (1) prediabetes; (2) lipid abnormalities; (3) elevated blood pressure. It is defined as occurring if any cardiometabolic abnormality has a reversal outcome at 12th month of study phrase.
  Reversal of cardiometabolic abnormalities is defined as: at 12th month of study phrase, at least one of the following status changed from abnormal at baseline to normal:
  i. Prediabetes; ii. Lipid abnormalities; iii. Elevated blood pressure.
Change in body fat (%) | From baseline to month 3
  Body fat(%) will be directly derived from non-invasive DEX body composition analyser, assessed by professional operator.
Change in the total score of the Wechsler Intelligence Scale for Children | From baseline to month 3
  Professionally trained and certified physicians will assess participants using the Wechsler Intelligence Scale for Children at baseline and at month 3 of the study, respectively, to obtain the total score of the scale (continuous variable outcome).
Change in body weight | From baseline to month 3
  Body weight is measured according to the Physical Fitness and Health Surveillance of Chinese School Students by trained, certified study staff. It is measured to the nearest 0.1 kg.
Change in body weight | From baseline to month 12
  Body weight is measured according to the Physical Fitness and Health Surveillance of Chinese School Students by trained, certified study staff. It is measured to the nearest 0.1 kg.
Change in waist circumference | From baseline to month 3
  Waist circumference is measured to the nearest 0.1 cm using a constant tension tape around the waist at 1 cm below the navel as the subject exhaled. It is calculated as the average value of two measurements.
Change in waist circumference | From baseline to month 12
  Waist circumference is measured to the nearest 0.1 cm using a constant tension tape around the waist at 1 cm below the navel as the subject exhaled. It is calculated as the average value of two measurements.
Change in fibroblast growth factor 21 (FGF-21) | From baseline to month 3
  FGF-21 will be measured by enzyme-linked immunosorbent assays (R&D Systems, Inc. USA), using fasting serum samples at baseline and month 3 after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China